CLINICAL TRIAL: NCT04276987
Title: A Pilot Clinical Study on Aerosol Inhalation of the Exosomes Derived From Allogenic Adipose Mesenchymal Stem Cells in the Treatment of Severe Patients With Novel Coronavirus Pneumonia
Brief Title: A Pilot Clinical Study on Inhalation of Mesenchymal Stem Cells Exosomes Treating Severe Novel Coronavirus Pneumonia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Collaborators: Shanghai Public Health Clinical Center (Other Government); Wuhan Jinyintan Hospital, Wuhan, China (Unknown); Shanghai AbelZeta Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MEXCOVID
Record Dates: First submitted 2020-02-16; First posted 2020-02-19 (Actual); Last update posted 2020-09-07 (Actual); Status verified 2020-09

CONDITIONS: Coronavirus
Keywords: mesenchymal stem cells; exosome; nebulization; SARS-CoV-2; novel coronavirus pneumonia
MeSH Terms: conditions — Coronavirus Infections

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MSCs-derived Exosomes Treatment Group (Experimental): Conventional treatment and aerosol inhalation of MSCs-derived exosomes treatment participants will receive conventional treatment and 5 times aerosol inhalation of MSCs-derived exosomes (2.0*10E8 nano vesicles/3 ml at Day 1, Day 2, Day 3, Day 4, Day 5).
  Interventions: Biological: MSCs-derived exosomes

INTERVENTIONS:
Biological: MSCs-derived exosomes — 5 times aerosol inhalation of MSCs-derived exosomes (2.0*10E8 nano vesicles/3 ml at Day 1, Day 2, Day 3, Day 4, Day 5).

SUMMARY:
In December 2019, a novel coronavirus infectious disease characterized by acute respiratory impairment due to severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) broke out in Wuhan city of Hubei province in China. So far no specific antiviral therapy can be available for patients with SARS-CoV-2 infection. Although symptomatic and supportive care, even with mechanical ventilation or extracorporeal membrane oxygenation (ECMO), are strongly recommended for severe infected individuals, those with advancing age and co-morbidities such as diabetes and heart disease remain to be at high risk for adverse outcomes. This pilot clinical trial will be performed to explore the safety and efficiency of aerosol inhalation of the exosomes derived from allogenic adipose mesenchymal stem cells (MSCs-Exo) in severe patients with novel coronavirus pneumonia (NCP).

DETAILED DESCRIPTION:
Since December 2019, SARS-CoV-2 infection has become a worldwide urgent public health event, especially in China. As of February 13, 2020, over 63,000 cases have been confirmed with over 10,200 severe cases in mainland of China. There is currently no vaccine or specific antiviral treatment existing for SARS-CoV-2 infection. Although symptomatic and supportive care are recommended for severe infected individuals, those with advancing age and co-morbidities such as diabetes and heart disease remain to be at high risk for adverse outcomes, with mortality of ~10%. Therefore, it is urgent to find a safe and effective therapeutic approach to patients with severe coronavirus disease-19(COVID-19) characterized by an severe acute respiratory impairment.

Experimental studies have demonstrated that mesenchymal stem cells (MSCs) or their exosomes (MSCs-Exo) significantly reduced lung inflammation and pathological impairment resulting from different types of lung injury. In addition, macrophage phagocytosis, bacterial killing and outcome are improved. It is highly likely that MSCs-Exo have the same therapeutic effect on inoculation pneumonia as MSCs themselves.

Although human bone marrow MSCs have been safely administered in patients with ARDS and septic shock (phase I/II trials), it seems safer to deliver MSCs-Exo rather than live MSCs. The intravenous administration of MSCs may result in aggregating or clumping in the injured microcirculation and carries the risk of mutagenicity and oncogenicity, which do not exist by treating with nebulized MSCs-Exo. Another advantage of MSCs-Exo over MSCs is the possibility of storing them for several weeks/months allowing their safe transportation and delayed therapeutic use.

The purpose of this single-arm design, open label, combined interventional clinical trial, therefore, is to explore the safety and efficiency of aerosol inhalation of the exosomes derived from allogenic adipose mesenchymal stem cells (MSCs-Exo) in the treatment of severe patients hospitalized with novel coronavirus pneumonia (NCP).

ELIGIBILITY:
Inclusion Criteria:

1.Willingness of study participant to accept this treatment arm, and signed informed consent; 2.Male or female, aged at 18 years (including) to 75 years old; 3.Patients with confirmed novel coronavirus pneumonia; 4.Confirmation of SARS-CoV-2 infection by reverse-transcription polymerase chain reaction (RT-PCR) from respiratory tract or blood specimens; 5.Diagnostic criteria of "Severe" or " Critical":

1. Severe, comply with any of the following:

   1. Respiratory distress, Respiratory rate (RR) ≥ 30 times/min
   2. Pulse oxygen saturation (SpO2) at rest ≤ 93%
   3. Partial pressure of oxygen/fraction of inspired oxygen (PaO2/FiO2) ≤ 300mmHg
2. Critical, comply with any of the following:

   1. Respiratory failure, and requirement for mechanical ventilation
   2. Shock
   3. Other organ failure and requirement for ICU monitoring

Exclusion Criteria:

1. Allergic or hypersensitive to any of the ingredients;
2. Pneumonia caused by bacteria, mycoplasma, chlamydia, legionella, fungi or other viruses;
3. Obstructive HABP/VABP induced by lung cancer or other known causes;
4. Carcinoid syndrome;
5. History of long-term use of immunosuppressive agents;
6. History of epilepsy and requirement for continuous anticonvulsant treatment or anticonvulsant treatment received within the last 3 years;
7. History of severe chronic respiratory disease and requirement for long-term oxygen therapy;
8. Undergoing hemodialysis or peritoneal dialysis;
9. Estimated or actual rate of creatinine clearance < 15 ml/min;
10. History of moderate and severe liver disease (Child-Pugh score >12);
11. Expectation of receiving any of following medications during the study:

    1. Receiving continuous valproic acid or sodium valproate within the first 2 weeks prior to screening
    2. Receiving 5-transtryptamine reuptake inhibitors, tricyclic antidepressants, 5-HT1 receptor agonists or monoamine oxidase inhibitors within the first 2 weeks prior to screening
12. Incapable of understanding study protocol;
13. History of deep venous thrombosis or pulmonary embolism within the last 3 years;
14. Undergoing ECMO or high-frequency oscillatory ventilation support;
15. HIV, hepatitis virus, or syphilis infection;
16. Period of pregnancy or lactation, or planned pregnancy within 6 months;
17. Any condition of unsuitable for the study determined by investigators.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2020-02-15 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
Adverse reaction (AE) and severe adverse reaction (SAE) | Up to 28 days
  Safety evaluation within 28 days after first treatment, including frequency of adverse reaction (AE) and severe adverse reaction (SAE)
Time to clinical improvement (TTIC) | Up to 28 days
  Efficiency evaluation within 28 days, including time to clinical improvement (TTIC)

SECONDARY OUTCOMES:
Number of patients weaning from mechanical ventilation | Up to 28 days
  Number of patients weaning from mechanical ventilation within 28 days
Duration (days) of ICU monitoring | Up to 28 days
  Duration (days) of ICU monitoring within 28 days
Duration (days) of vasoactive agents usage | Up to 28 days
  Duration (days) of vasoactive agents using within 28 days
Duration (days) of mechanical ventilation supply | Up to 28 days
  Duration (days) of mechanical ventilation supply among survivors
Number of patients with improved organ failure | Up to 28 days
  Number of patients with improved organ failure within 28 days, including cardiovascular system, coagulation system, liver, kidney and other extra-pulmonary organs
Rate of mortality | Up to 28 days
  Rate of mortality within 28 days

OTHER OUTCOMES:
Sequential organ failure assessment (SOFA) score | Every day for 28 days
  Records of daily sequential organ failure assessment (SOFA) score (From 0 to 24 points, higher scores mean a worse outcome)
Lymphocyte Count (10E9/L) | Day0, Day3, Day7, Day14, Day21, Day28, indicated time points can be added if available
  Records of Blood routine test
C-reactive protein (CRP) (mg/L) | Day0, Day3, Day7, Day14, Day21, Day28, indicated time points can be added if available
Lactate dehydrogenase (U/L) | Day0, Day3, Day7, Day14, Day21, Day28, indicated time points can be added if available
D-dimer (mg/L) | Day0, Day3, Day7, Day14, Day21, Day28, indicated time points can be added if available
  Coagulation function
pro-type B natriuretic peptide (pro-BNP) (pg/ml) | Day0, Day3, Day7, Day14, Day21, Day28, indicated time points can be added if available
  Records of heart failure
IL-1β (pg/ml) | Day0, Day3, Day7, Day14, Day21, Day28, indicated time points can be added if available
  Record of serum cytokine
IL-2R (ng/L) | Day0, Day3, Day7, Day14, Day21, Day28, indicated time points can be added if available
  Record of serum cytokine
IL-6 (ng/L) | Day0, Day3, Day7, Day14, Day21, Day28, indicated time points can be added if available
  Record of serum cytokine
IL-8 (ng/L) | Day0, Day3, Day7, Day14, Day21, Day28, indicated time points can be added if available
  Record of serum cytokine
Chest imaging | Day0, Day3, Day7, Day14, Day21, Day28, indicated time points can be added if available
  Computed tomography or X-ray
Time to SARS-CoV-2 RT-PCR negativity | Up to 28 days
  Time to SARS-CoV-2 RT-PCR negativity in respiratory tract specimens

CONTACTS AND LOCATIONS:
Overall Officials: Jie-ming Qu, MD.,PhD., Principal Investigator — Ruijin Hospital, Medical School of Shanghai Jiaotong University Shanghai, China
Locations (1):
- Ruijin Hospital Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Starting 6 months after publication

REFERENCES:
- [Derived] Zhu YG, Shi MM, Monsel A, Dai CX, Dong X, Shen H, Li SK, Chang J, Xu CL, Li P, Wang J, Shen MP, Ren CJ, Chen DC, Qu JM. Nebulized exosomes derived from allogenic adipose tissue mesenchymal stromal cells in patients with severe COVID-19: a pilot study. Stem Cell Res Ther. 2022 May 26;13(1):220. doi: 10.1186/s13287-022-02900-5. PMID 35619189